CLINICAL TRIAL: NCT06848868
Title: Flexible Ureterorenoscopy for Surveillance of Upper Tract Urothelial Carcinoma-A Pilot Study
Brief Title: Ambulatory Flexible URS for UTUC Surveillance
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong, Ho Ming Chris, Resident Doctor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB/REC 2024.432
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: UTUC; Upper tract urothelial carcinoma; Ureterorenoscopy; Flexible ureterorenoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory flexible ureterorenoscopy (Experimental)
  Interventions: Procedure: Ambulatory flexible ureterorenoscopy

INTERVENTIONS:
Procedure: Ambulatory flexible ureterorenoscopy — Ambulatory flexible ureterorenoscopy (experimental)

SUMMARY:
This is a a prospective single-arm pilot study to investigate the safety and feasibility of flexible ureteroscopy under local anaesthesia. All consecutive patients who have undergone kidney-sparing surgery for managing upper tract urothelial carcinoma will be screened for study eligibility. The primary outcome is the procedural technical success rate. Secondary outcomes include the 30-day complication rate following flexible ureteroscopy, readmission rates, cost analysis, and patient-reported outcomes. Ureterorenoscopy will be conducted in the recruited patients under local anaesthesia in the ambulatory urology centre. Procedural details, technical success rates, adverse events and patient reported outcomes will be documented. The anticipated risks of this intervention are not expected to exceed those associated with the standard of care, that is ureterorenoscopy under anaesthesia. This pilot study aims to recruit a total of 10 subjects to assess the safety and feasibility of flexible ureterorenoscopy in an ambulatory care setting.

DETAILED DESCRIPTION:
The study is designed to examine the safety and feasibility to conduct surveillance flexible ureteroscopy of the upper urinary tract under local anaesthesia in an ambulatory care setting.

The study is intended to identify patients who have undergone kidney-sparing surgery for upper tract urothelial carcinoma with need of surveillance of the upper urinary tract.

Prior to procedure, mid-stream or catheterised urine samples will be collected two weeks beforehand. To ensure a sterile urinary tract, asymptomatic bacteriuria will be treated with antibiotics tailored to the urine culture results, or with broad spectrum antibiotics. Anti-platelet or anticoagulation medications will be discontinued in accordance with local guidelines prior to the operation.

Procedures will be conducted by experienced urology specialists.The procedure will commence with the patient in a supine position, followed by the administration of transurethral lidocaine jelly five minutes prior to the procedure - either in room temperature or chilled preparation. Additional intravenous sedative medication prior to the endoscopic examination will be optional.

Initially, a flexible cystoscope will be introduced to examine the bladder and ureteric orifices, and a lower tract surveillance will be performed. In cases without a pre- existing ureteric double J stent, the ureteric orifice may be cannulated with a guidewire, followed by the introduction of a flexible ureteroscope, either alongside or railroading the guidewire.

The decision to use a guidewire in cases with tight ureteric orifices will be made by the operating urologist. If a ureteric double J stent is in situ, it will be retrieved using foreign body forceps with a flexible cystoscope, and a guidewire will be used for the stent exchange, then the flexible ureteroscope will be introduced alongside or railroading the guidewire.

The choice of ureteroscope will be left to the operating urologist's discretion. The procedure will either be performed with a reusable or a disposable fURS. The fURS will be inserted to the renal pelvis by direct vision. A complete renoscopy for the tip of the fURS deflecting to the different calyces will be performed. After renoscopy, the fURS will be carefully and slowly withdrawn. Saline irrigation through the instrumental channel will continually take place to ensure visibility of the lumen. During withdrawal, the ureter will be inspected, until the fURS is retrieved through the ureteric orifice. During renoscopic and ureteroscopic examination, findings will be documents in a pre-specified electornic form. Any suspicious mucosal lesion may be biopsied, subject to the operating urologist's judgment. A circulating nurse will monitor the patient's blood pressure, pulse, and pulse oximetry throughout the procedure. Should the patient experience intolerable discomfort or significant derangement in vital signs, the procedure will be immediately ceased.

Post-procedure, patients will be observed in the observation are of the ambulatory centre. Vital signs including blood pressure, pulse, oxygen saturation, and temperature will be monitored. Patients who do not require an indwelling urinary catheter will be encouraged to void, and their post-void residual urine volume will be recorded. Discharge from the ambulatory unit will be authorized only if the patient's vital signs remain stable and they demonstrate adequate voiding.

Upon discharge, all baseline characteristics and peri-procedural complications will be meticulously recorded in a designated electronic form. Complications will be graded using the Clavien-Dindo classification, and electronic records will be reviewed for up to 30 days post-procedure to document any instances of hospital attendance and the reasons thereof. i.e., ureterorenoscopy under anesthesia in an operating theatre. However, should any suspected ureteric injury or avulsion occur-a risk also inherent in standard procedures-the ureterorenoscopy will be halted, a double J stent will be placed via the guidewire, and the patient will be admitted to an inpatient ward for further monitoring and management.

The participants will be continually monitored if they suffer from any adverse event, till resolution of the event. All patients who experience an adverse event (AE) will be evaluated at appropriate time intervals until the event resolves or stabilizes. At the conclusion of the study, the investigator will assess unresolved AE and determine if additional follow-up is warranted based on clinical assessment.

Collection of Serious adverse event (SAE) information will begin at the time the patient signs the informed consent and continue through screen failure, end of study follow-up, or safety follow-up if the condition is not resolved or stabilized All SAE must be followed with appropriate medical management until resolved or until progression has been stabilized.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Capable of giving informed consent
3. Having undergone an kidney-sparing surgery (endoscopic operation or segmental ureterectomy)

Exclusion Criteria:

1. Allergy to transurethral lidocaine jelly
2. On anticoagulation or anti-platelet medication with contraindications for cessation prior to the procedure
3. Structural abnormalities in the upper urinary tract on the intended side of examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical success of the flexible ureterorenoscopy | Perioperative/Periprocedural
  Technical success of the flexible ureterorenoscopy, defined as complete visualisation of all renal calyces and the entire course of the ureter.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be shared upon contacting the principal investigator

REFERENCES:
- [Background] Jain K, Blachman-Braun R, Jain E, Eng A, Peters B, Patel P. Ureteroscopy under conscious sedation: A proof-of-concept study. Can Urol Assoc J. 2022 Sep;16(9):E461-E467. doi: 10.5489/cuaj.7750. PMID 35426786
- [Background] Peng Y, Wang L, Jin J, Jiang Y, Xu Q, Yang L, Liu J. Flexible ureteroscopy under local anesthesia for stone management: initial exploration and two-year experience. Postgrad Med. 2023 Sep;135(7):755-762. doi: 10.1080/00325481.2023.2265991. Epub 2023 Oct 24. PMID 37773585
- [Background] Villa L, Cloutier J, Letendre J, Ploumidis A, Salonia A, Cornu JN, Montorsi F, Traxer O. Early repeated ureteroscopy within 6-8 weeks after a primary endoscopic treatment in patients with upper tract urothelial cell carcinoma: preliminary findings. World J Urol. 2016 Sep;34(9):1201-6. doi: 10.1007/s00345-015-1753-7. Epub 2015 Dec 23. PMID 26699629
- [Background] Cybulski PA, Joo H, Honey RJ. Ureteroscopy: anesthetic considerations. Urol Clin North Am. 2004 Feb;31(1):43-7, viii. doi: 10.1016/S0094-0143(03)00087-9. PMID 15040400
- [Background] Zganjar AJ, Thiel DD, Lyon TD. Diagnosis, workup, and risk stratification of upper tract urothelial carcinoma. Transl Androl Urol. 2023 Sep 30;12(9):1456-1468. doi: 10.21037/tau-23-45. Epub 2023 Aug 4. PMID 37814699
- [Background] Pandolfo SD, Cilio S, Aveta A, Wu Z, Cerrato C, Napolitano L, Lasorsa F, Lucarelli G, Verze P, Siracusano S, Quattrone C, Ferro M, Bologna E, Campi R, Del Giudice F, Bertolo R, Amparore D, Palumbo S, Manfredi C, Autorino R. Upper Tract Urothelial Cancer: Guideline of Guidelines. Cancers (Basel). 2024 Mar 11;16(6):1115. doi: 10.3390/cancers16061115. PMID 38539450
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303